CLINICAL TRIAL: NCT02622152
Title: Right Lateral Positioning of Postoperative Pediatric Cardiac Surgery: Effect on Arterial Oxygenation, Respiratory Mechanics, Hemodynamics, and Adverse Events
Brief Title: Right Lateral Positioning of Postoperative Pediatric Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB0000871200
Record Dates: First submitted 2015-11-28; First posted 2015-12-04 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Heart Defects, Congenital
Keywords: Right lateral; Oxygenation; Cardiac; Congenital; Pediatric; Postoperative
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right lateral position group (Active Comparator): After weaning from mechanical ventilation in the postoperative Intensive Care Unit (ICU patient underwent Repositioning the patients for 30 minutes period on the supine position Repositioning the patients for 30 minutes period on the left lateral position Repositioning the patients for two-hours period on the right lateral position This period of repositioning in both groups repeated during the period of ICU stay
  Interventions: Procedure: Right lateral position (2 hours); Procedure: Left lateral position (30 minutes); Procedure: Supine position (30 minutes)
- Routine hospital care group (Active Comparator): After weaning from mechanical ventilation in the postoperative Intensive Care Unit (ICU patient underwent Repositioning the patients for two-hours period on supine position Repositioning the patients for two-hours period on the left lateral position Repositioning the patients for two-hours period on the right lateral position This period of repositioning in both groups repeated during the period of ICU stay
  Interventions: Procedure: Right lateral position (2 hours); Procedure: Left lateral position (2 hours); Procedure: Supine position (2 hours)

INTERVENTIONS:
Procedure: Right lateral position (2 hours) — Repositioning the patients for two-hours period on the right lateral position
Procedure: Left lateral position (30 minutes) — Repositioning the patients for 30 minutes period on the left lateral position
  Arms: Right lateral position group
Procedure: Supine position (30 minutes) — Repositioning the patients for 30 minutes period on the supine position
  Arms: Right lateral position group
Procedure: Left lateral position (2 hours) — Repositioning the patients for two-hours period on the left lateral position
  Arms: Routine hospital care group
Procedure: Supine position (2 hours) — Repositioning the patients for two-hours period on supine position
  Arms: Routine hospital care group

SUMMARY:
Directly following cardiac surgery for congenital heart disease; patients are not receiving routine turning every two hours to prevent pressure ulcers, because a negative influence on hemodynamic parameters is assumed. Investigators have suggested that lateral position may have clinically significant effects on oxygenation in cardiac surgery patients.

DETAILED DESCRIPTION:
Sixty pediatric congenital heart disease patients were randomly assigned to two equal intervention groups

ELIGIBILITY:
Inclusion Criteria:

* Age within 10 years with a cyanotic congenital heart disease
* Hemodynamic stability with no compromising arrhythmia
* No respiratory arrest
* Not connected with mechanical ventilation

Exclusion Criteria:

* Cyanotic congenital heart disease
* Hemodynamic instability

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-01-30 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Arterial oxygenation | Duration of Intensive Care Unit Admission after weaning from mechanical ventilation an expected average of 4 days
  The samples will be analyzed by a blood gas analyzer before and after changing position

SECONDARY OUTCOMES:
Blood pressure | Duration of Intensive Care Unit Admission after weaning from mechanical ventilation an expected average of 4 days
  Systolic, diastolic and mean blood pressure " mm Hg"
Heart rate | Duration of Intensive Care Unit Admission after weaning from mechanical ventilation an expected average of 4 days
  Heart rate "beats per minute"
Oxygen saturation | Duration of Intensive Care Unit Admission after weaning from mechanical ventilation an expected average of 4 days
  Oxygen saturation %
Respiratory rate | Duration of Intensive Care Unit Admission after weaning from mechanical ventilation an expected average of 4 days
  Respiratory rate "rate per minute"

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, MD, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided